CLINICAL TRIAL: NCT05648396
Title: Japan Multicentre FFRangio Outcomes Registry
Brief Title: Japan FFRangio Clinical Outcomes Study
Status: Active, not recruiting | Type: Observational
Sponsor: Rabin Medical Center (Other)
Collaborators: Gifu Heart Center (Other); Fukuoka Sanno Hospital (Unknown); Saga-ken Medical Center Koseikan (Unknown); Sakakibara Heart Institute (Other); Fukuyama Cardiovascular Hospital (Unknown); Ichinomiya-Nishi Hospital (Unknown)
Responsible Party: Principal Investigator, Guy Witberg, Consultant inteventional cardiologist, Rabin Medical Center
Other Study IDs: RMC-12-2022
Record Dates: First submitted 2022-11-12; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Revascularization: Patients undergoing angiogram in which FFRangio is used to assess the physiologic significance of at least one coronary lesion, and based on this assessment are referred for coronary revascularization (PCI/CABG).
  Interventions: Other: FFRangio
- Deferral: Patients undergoing angiogram in which FFRangio is used to assess the physiologic significance of at least one coronary lesion, and based on this assessment are assigned to conservative management (optimal guidelines directed medical treatment).
  Interventions: Other: FFRangio

INTERVENTIONS:
Other: FFRangio — Assessing the physiologic significance of an intermediate coronary lesion/lesions using FFRangio - a non invasive method to calculate the fractional flow reserve (FFR) of the assessed lesion.

SUMMARY:
This study aims to collect data on clinical outcomes of real world patients undergoing FFRangio guided treatment for coronary artery disease in Japan and Israel through a retrospective multicentre registry.

DETAILED DESCRIPTION:
Background:

Visual assessment of the severity of coronary stenosis is known to have a poor diagnostic accuracy for identifying functionally significant lesion [1,2). The fractional flow reserve (FFR) is an index that quantifies the hemodynamic impact of a stenosis in an epicardial coronary artery. It is defined as the ratio of hyperemic myocardial flow in the presence of stenosis to the hyperemic flow in its absence, and is obtained by measuring the distal coronary pressure and the aortic pressure, respectively, using a pressure-measuring guidewire during maximal hyperemia [2,3]. Clinical outcome studies have shown that medical therapy should be preferred for non-hemodynamically significant lesions (FFR>0.80), and coronary revascularization should be considered in cases of significant functional stenosis (FFR≤0.80) [4-11]. Accordingly, both American and European revascularization guidelines recommend using FFR to guide coronary revascularization, especially in stable coronary artery disease patients [12,13]. In spite of these recommendations, the utilization of FFR in clinical practice remains low [14]. Recently, methods to calculate angiogram based FFR (abFFR) (without the need for pressure wires or induction of maximal coronary hyperemia) have become available. A meta-analysis of 14 studies examining various abFFR technologies ( total of 1,842 lesions), reported a sensitivity of 89%, specificity of 90%, and a C-statistic of 0.84 compared to wire based FFR (wbFFR) [15], highlighting the potential for abFFR technologies to facilitate the integration of physiologic assessment into daily cathlab practice. The FFRangioTM system (CathWorks, Kfar-Saba, Israel; Figure 1), is an angiogram-derived FFR technology that has shown excellent diagnostic performance (overall accuracy 92.6%) when compared to wire based FFR in a large pooled cohort of individual patients data from 5 individual studies (588 patients, 700 lesions) [16]. FFRangio has already received FDA 510(k) clearance for clinical use as a stand-alone technology without the need for concurrent wire based FFR measurement [17]. FFRangio has been in clinical use in Japan since 2019, but there is very limited data on the clinical outcomes of FFRangio guided treatment.

Recently, the first study examining the outcomes of FFRangio guided treatment for patients undergoing angiography for suspected coronary artery disease has reported excellent 1 year results for both FFRangio guided revascularization as well as deferral [18], but more data is needed to more appropriately assess the technology in real world patients.

The aim of this multicenter registry is to expand the evidence base on outcomes of FFRangio guided treatment for coronary artery disease, focusing on outcomes of Japanese patients.

Methods:

A retrospective, multicenter registry of consecutive patients in whom FFRangio is used to assess the physiologic significance of at least 1 coronary lesion and guide the treatment decisions .

Inclusion criteria:

• Patients undergoing coronary angiogram for a clinical indication, for whom FFRangio is used to assess the physiologic significance of at least 1 coronary lesion and guide the treatment decisions.

Exclusion criteria:

* Culprit lesion of a STEMI (patients undergoing PCI for non-culprit lesions can be included if the culprit lesion has been successfully treated prior to the non-culprit PCI
* Presence of significant (moderate+) valvular heart disease
* Chronic total occlusion in one of the coronary arteries
* Isolated significant left main disease
* Prior coronary artery bypass graft surgery
* Clinical presentation of cardiogenic shock or severe LV dysfunction
* Coronary anomalies

Endpoints

Primary endpoint:

• composite of all cause death/myocardial infarction(MI)/repeat revascularization(RR) at 1 year follow up.

Secondary endpoints:

* The individual components of the primary endpoint
* Cardiovascular (CV) death
* Urgent RR (performed as an inpatient during an admission for ACS).
* Target vessel RR
* Target lesion RR
* Target vessel MI
* Target lesion MI

Timing of follow up:

Six and 12 months post procedure (primary analysis will include 1 year data) and yearly follow up thereafter up to 5 years.

Ascertainment and adjudications of clinical events The clinical endpoints events will be identified by the participating centres through the patients' electronic medical record and will be further verified, when possible, by interviews conducted during in person/virtual outpatient clinic visits and/or telephone follow up.

Sample size Our aim is to include up to 10 high volume FFRangio centres from Japan and Israel with a goal of reaching a sample size of at least 1,500 patients.

Ethical aspects The study will be approved by the local institutional review boards at each participating centre. Since there is no intervention in the clinical care given to the patient, waiver of the need for patient's informed consent will besought from the IRB/EC.

If participating investigators come by patients' personal information ( information on living individuals that can be used to specific individuals by name, date of birth or other description), such information shall be treated and protected under strict confidentiality. Further more participating investigators shall conduct this research in accordance with ethical principles on the Declaration of Helsinki.

Expected time frame Initiation of registry: Q4 2022 Expected data collection for 1,500 patients: Q2 2023 Initial data analysis: Q3 2023 (median follow up of 6 months for a sample size of 1,500 patients )

ELIGIBILITY:
Inclusion criteria:

• Patients undergoing coronary angiogram for a clinical indication, for whom FFRangio is used to assess the physiologic significance of at least 1 coronary lesion and guide the treatment decisions.

Exclusion criteria:

* Culprit lesion of a STEMI (patients undergoing PCI for non-culprit lesions can be included if the culprit lesion has been successfully treated prior to the non-culprit PCI
* Presence of significant (moderate+) valvular heart disease
* Chronic total occlusion in one of the coronary arteries
* Isolated significant left main disease
* Prior coronary artery bypass graft surgery
* Clinical presentation of cardiogenic shock or severe LV dysfunction
* Coronary anomalies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all comers patients undergoing coronary angiogram, in which FFRangio is used to assess the physiologic significance of at least one coronary lesion.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
composite of Cardio-Vascular(CV) mortality/Myocardial infarction (MI)/Repeat revascularization | 1 year
  Composite of CV mortality/MI/Repeat revascularization

SECONDARY OUTCOMES:
Overall death | 1 year
  Death due to any cause
Cardio Vascular death | 1 year
  Death due to a Cardiovascular cause
MyocardiaI infarction (MI) | 1 year
  Defined by the universal definition of MI
Repeat revascularization | 1 year
  Any revascularization procedure
Urgent repeat revascularization | 1 year
  Any revascularization procedure performed urgently (i.e as an inpatient with an indication of acute coronary syndrome)
target vessel repeat revascularization | 1 year
  Any revascularization procedure involving the target vessel assessed during the index procedure
Target lesion repeat revascularization | 1 year
  Any revascularization procedure involving the target lesion assessed during the index procedure
Target vessel MI | 1 year
  Any MI related to target vessel assessed during the index procedure
Target lesion MI | 1 year
  Any MI related to target lesion assessed during the index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Guy Witberg, MD, MPH, Principal Investigator — Rabin Medical Centre
Locations (1):
- Rabin Medical Centre, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witberg G, Kikuta Y, Dan K, Matsumura M, Maehara A, Tanigaki T, Yokoi H, Hikichi Y, Nanasato M, Miura K, Sato K, Taniguchi M, Goto K, Haruta S, Levi A, Otake H, Fearon WF, Matsuo H, Kornowski R, Takebayashi H. Mid-term clinical outcomes of FFRangio guided treatment for coronary artery disease: Insights from an international multicentre registry. Cardiovasc Revasc Med. 2026 Jan 23:S1553-8389(26)00013-8. doi: 10.1016/j.carrev.2026.01.012. Online ahead of print. PMID 41620337
- [Derived] Dan K, Witberg G, Itabashi F, Maeda T, Kikuta Y, Okabe K, Tanigaki T, Nanasato M, Hikichi Y, Yokoi H, Kornowski R, Matsuo H. Comparison of angiogram-based physiological assessment system sizing tool and intravascular ultrasound imaging measurements. Cardiovasc Revasc Med. 2025 Sep;78:80-85. doi: 10.1016/j.carrev.2025.03.012. Epub 2025 Mar 18. PMID 40148172